CLINICAL TRIAL: NCT02468375
Title: A Multicenter Prospective Study for Patient Perception of Treatment Satisfaction After Switching to Mirabegron in Patients With Overactive Bladder Who Were Unsatisfied With Efficacy of Antimuscarinic Therapy or Adverse Event.
Brief Title: Prospective Study for Patient Perception of Treatment Satisfaction After Switching to Mirabegron in Patients With Overactive Bladder Who Were Unsatisfied With Efficacy of Antimuscarinic Therapy or Adverse Event.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-02-052
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2015-06

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mirabegron 50mg (Experimental): about 434 OAB patients intake mirabegrone 50mg/day for 12 weeks.
  Interventions: Drug: mirabegron 50mg

INTERVENTIONS:
Drug: mirabegron 50mg — 434 OAB patient intake mirabegron 50mg/day for 12 weeks.
  Other Names: Betamiga tablet

SUMMARY:
The purpose of this study is to measure the treatment satisfaction after switching to mirabegron in patient with Overactive Bladder(OAB) who were unsatisfied with efficacy of antimuscarinic therapy or adverse event.

Patient will take the mirabegron 50mg/day for 12 weeks, and the satisfation of the therapy will be measured with Treatment Satisfaction Questionnaire(TSQ), Global Response Assessment(GRA), OAB-q short form, OAB Symptom Score and Willingness to continue Questions.

ELIGIBILITY:
Inclusion Criteria:

<SCREENING>

1. over 20 years old, who has overactive bladder at least for 3 months.
2. total OABSS score over 3 points, and number 3 question score should be over 2 points.
3. if one of the criteria met,

1) efficacy : who are unsatisfied with antimuscarinics during the past 2 years. (should be treated at least 8 weeks) 2) adverse event(AE) : who are unsatisfied with antimuscarinics treatment due to AE(dry mouth, constipation, etc) 4.subject who can write voiding diary. 5.subject who can understand about the study and sign the informed concent form.

<BASELINE> Voiding Diary for 3 days

1. micturition 8/day
2. urgency 2/day

Exclusion Criteria:

<SCREENING>

1. subject has history or risk of acute urinary retension.
2. subject has prostate cancer.
3. subject has lower urinary tract obstruction and judge by investigator that the subject is not appropriate to participate in this study.
4. subject has a previous or current bladder tumor.
5. subject has significant stress incontinence or mixed incontinence where stress is the dominant factor.
6. prohibitied, permitted medication. 6-1. subject who has intake Alpha-blocker, Diabetes insipidus medication, PDE5 inhibitor(for BPH Tx), SSRI within 12weeks prior to Screening.

   6-2. subject who has started, stopped or changed the dose of 5-Alpha Reductase Inhibitors(5-ARI) within 4 weeks prior to Screening.

   6-3. Subject who currently intake Antimuscarinics, Antihistamines, Beta 2-adrenoreceptor agonist, loop diuretics,CYP2D6 substrates with narrow therapeutic index, CYP3A4 inducing agent, CYP 3A4 inhibitor, Antifungal agent, Antiarrythmic drugs.
7. subject who has Non-drug treatment including bladder training, pelvic floor muscle training within 12 weeks prior to Screening.
8. subject has severe hypertension which is defined as a sitting average systolic blood pressure over 180 mmHg, and/or diastolic blood pressure over 11 0mmHg.
9. pulse over 100 bpm or below 50 bpm.
10. subject has an indwelling catheter or practices intermittent self-catheterization.
11. subject who had surgery which can influence urinary track function (ex, TURP, Laser treatment,etc.).
12. subject who had complication of urinary tract infection, urinary stone, interstitial cystitis, or recurrent UTI history.
13. subject has known or suspected hypersensitivity to Beta 3 adrenalin receptor agonist.
14. subject has clinically significant cardiovascular diseases hepatic diseases renal diseases immunization diseases lung diseases and cancer.
15. subject who has planed pregnency, breast feeding during clinical trial period.

<BASELINE> voiding volume over 3000ml per day. post voiding residual volume over 200ml

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2015-06; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfation Questionnaire | at the end of the treatment( 12weeks)

SECONDARY OUTCOMES:
micturtion change | 4weeks, 12weeks
urgency change | 4weeks, 12weeks
incontinence change | 4weeks. 12weeks
OABq-SF score change | 4weeks, 12weeks
OABSS score change | 4weeks, 12weeks
Global Response Assessment(GRA) score change | 4weeks, 12weeks
Willingness to continue Questions | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea